CLINICAL TRIAL: NCT04656626
Title: Brief Mindfulness Based Intervention for Front-Line Medical Staff in the COVID19 Pandemic to Improve Psychological Wellbeing, a Randomized Controlled Multicenter Trial
Brief Title: Brief Mindfulness Based Intervention to Improve Psychological Wellbeing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imam Abdulrahman Bin Faisal University (Other)
Responsible Party: Principal Investigator, Amani M AlQurni, Assistant Professor - Family Medicine, Imam Abdulrahman Bin Faisal University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: Mindfullness during a pandemic
Record Dates: First submitted 2020-12-04; First posted 2020-12-07 (Actual); Last update posted 2020-12-10 (Actual); Status verified 2020-12

CONDITIONS: Stress, Psychological
MeSH Terms: conditions — Stress, Psychological | interventions — Autogenic Training

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: masking/ blindness was programmed in the system/website that was developed for this study; the participants, those administering the interventions, and those assessing the outcomes were blinded to group assignment.
  the system/ website For the sack of this study a new system was developed to be used for data collection. The system was designed as an electronic questioner with audio clips that is sent automatically to the participants' email and phones, where each participant receives their own special link.
  the participants after responding to the pre intervention link will be automatically randomized by the system/website to intervention or control group.
  the whole data collection and intervention process is automatic, virtual and blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COVID19 Frontline Health Care Providers recieving mindfulness intervention (Experimental): This arm will receive mindfulness audios (randomized and double blinded)
  Interventions: Behavioral: brief mindfulness based intervention
- COVID19 Frontline Health Care Providers receiving progressive muscle relaxation (Placebo Comparator): This arm will receive progressive muscle relaxation audios (randomized and double blinded)
  Interventions: Behavioral: Progressive muscle relaxation

INTERVENTIONS:
Behavioral: brief mindfulness based intervention — The 20 minute daily mindfulness sessions for 2 weeks consist of the following guided meditation practices: 1. Bring your attention to a primary object of focus 2. Maintain a moment-moment awareness 3. When your mind naturally drifts into thinking (mind wandering); just notice you are thinking, and then bring your attention back to your object of focus 4. When a strong sensation arises, again, notice the sensation or emotion and return to your breath. 5. As you gain confidence, you may practice maintaining this focus while observing thoughts flowing through your mind or sensations in your body while showing no concern for the content 6. You may even label your thoughts 7. Thank yourself for your efforts and for taking this time.
  Arms: COVID19 Frontline Health Care Providers recieving mindfulness intervention
Behavioral: Progressive muscle relaxation — Control group:
  Control group will be given an mp3 audio recording of a 20-minutes of progressive muscle relaxation will be sent directly as SMS messages and emails to be heard by the participants through their personal device of their choice, such as a smart phone.
  Arms: COVID19 Frontline Health Care Providers receiving progressive muscle relaxation

SUMMARY:
our aim is to evaluate the effectiveness of virtual brief mindfulness based interventions on psychological wellbeing, resiliency, and anxiety of frontline HCP to cope for (COVID19) stressors

DETAILED DESCRIPTION:
Our specific objectives are: To measure frontline HCP's level of anxiety, resilience, and how mindfulness based interventions affect anxiety and psychological resilience of HCP.

ELIGIBILITY:
Inclusion Criteria:

* COVID19 frontline health care providers namely, physicians, nurses and respiratory therapist at 2 main hospitals in the eastern province of KSA

Exclusion Criteria:

1. History of psychotic disorder,
2. Substance abuse or dependence within the last 6 months
3. Current severe neurotic disorder, severe depression or severe anxiety.
4. Concurrent psychotherapy.
5. Significant personality disorder

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2020-07-07 (Actual); Primary Completion 2020-07-21 (Actual); Study Completion 2020-09-05 (Actual)

PRIMARY OUTCOMES:
reduction of anxiety symptom severity | 14 days
  assessed using the (state trait anxiety-7 Item Scale); ranged from 10-40, higher score indicate more anxiety
change in the level of psychological resilience | 14 days
  assessed using the (Connor-Davidson Resilience Scale (CD-RISC)); score from 0-40, higher scores indicate more resilience

SECONDARY OUTCOMES:
mental wellbeing | 14days
  assessed by World Health Organization wellbeing scale; changed to percent score, the higher the better.
and functional status | 14 days
  12-Item Short Form survey

CONTACTS AND LOCATIONS:
Overall Officials: amani al-qurni, BOARD, Principal Investigator — IMAM ABDULRHMAN BIN FAISAL UNIVERSITY
Locations (1):
- Imam Abdulrahman Bin Faisal University, Dammam, Saudi Arabia

REFERENCES:
- [Background] Alzahrani AM, Hakami A, AlHadi A, Batais MA, Alrasheed AA, Almigbal TH. The interplay between mindfulness, depression, stress and academic performance in medical students: A Saudi perspective. PLoS One. 2020 Apr 3;15(4):e0231088. doi: 10.1371/journal.pone.0231088. eCollection 2020. PMID 32243468
- [Background] Lynn SJ, Barnes S, Deming A, Accardi M. Hypnosis, rumination, and depression: catalyzing attention and mindfulness-based treatments. Int J Clin Exp Hypn. 2010 Apr;58(2):202-21. doi: 10.1080/00207140903523244. PMID 20390691
- [Background] Lau MA, Bishop SR, Segal ZV, Buis T, Anderson ND, Carlson L, Shapiro S, Carmody J, Abbey S, Devins G. The Toronto Mindfulness Scale: development and validation. J Clin Psychol. 2006 Dec;62(12):1445-67. doi: 10.1002/jclp.20326. PMID 17019673
- [Background] Brooks SK, Gerada C, Chalder T. Review of literature on the mental health of doctors: are specialist services needed? J Ment Health. 2011 Apr;20(2):146-56. doi: 10.3109/09638237.2010.541300. Epub 2011 Jan 28. PMID 21275504
- [Background] Carmody J, Baer RA. Relationships between mindfulness practice and levels of mindfulness, medical and psychological symptoms and well-being in a mindfulness-based stress reduction program. J Behav Med. 2008 Feb;31(1):23-33. doi: 10.1007/s10865-007-9130-7. Epub 2007 Sep 25. PMID 17899351

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-05-05): https://cdn.clinicaltrials.gov/large-docs/26/NCT04656626/Prot_SAP_000.pdf
  • Informed Consent Form (2020-05-01): https://cdn.clinicaltrials.gov/large-docs/26/NCT04656626/ICF_001.pdf